CLINICAL TRIAL: NCT05276596
Title: Evaluation of the Early Use of Norepinephrine in Major Abdominal Surgery on Postoperative Organ Dysfunction
Acronym: EPON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2021_843_0060
Record Dates: First submitted 2022-03-03; First posted 2022-03-11 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Norepinephrine; Hypotension; Anesthesiology; Major Abdominal Surgery
Keywords: norepinephrine; ephedrine; Hypotension; anesthesiology; major abdominal surgery; Clavien Dindo score
MeSH Terms: conditions — Hypotension | interventions — Ephedrine; Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The first anesthetic post-induction hypotension will be managed by intravenous injection of ephedrine (dilution: 3 mg / ml) at a dose of 6 mg (i.e. 2 ml). Any subsequent hypotension will be treated with ephedrine until injection of a total dose of 30 mg. Thereafter, if a new arterial hypotension occurs, we will pass to the administration of noradrenaline in intravenous injection using an electric syringe pump, at the dilution of 0.016 mg / ml, posology adapted to the objectives. blood pressure.
  Interventions: Drug: Ephedrine
- Test group (Experimental): Immediately use of norepinephrine by intravenous injection using an electric syringe pump, at a dilution of 0.016 mg / ml, at the time of anesthetic induction and without waiting the 1st possible arterial hypotension. Noradrenaline will be started at a dose of 0.48 mg / h and then adapted according to the blood pressure objectives.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Ephedrine — The control group will be taken care of according to the protocols in force. The first anesthetic post-induction hypotension will be managed by intravenous injection of ephedrine (dilution: 3 mg / ml) at a dose of 6 mg (i.e. 2 ml). Any subsequent hypotension will be treated with ephedrine until injection of a total dose of 30 mg. Thereafter, if a new arterial hypotension occurs, we will pass to the administration of noradrenaline in intravenous injection using an electric syringe pump, at the dilution of 0.016 mg / ml, posology adapted to the objectives. blood pressure.
  Arms: Control group
Drug: Norepinephrine — Immediately use of norepinephrine by intravenous injection using an electric syringe pump, at a dilution of 0.016 mg / ml, at the time of anesthetic induction and without waiting the 1st possible arterial hypotension. Noradrenaline will be started at a dose of 0.48 mg / h and then adapted according to the blood pressure objectives.
  Arms: Test group

SUMMARY:
Hemodynamic instability is frequent during surgery and intraoperative hypotension is associated with excess morbidity and excess mortality in high-risk patients. In major abdominal surgery the incidence of intraoperative hypotension remains high.

For the past few years, some teams have proposed evaluating norepinephrine as a first-line drug in the presence of hypotension or even before hypotension occurs Thus in obstetrics, the preventive use of norepinephrine for cesareans performed under spinal anesthesia was associated with a reduction in the incidence of hypotension per operative without deleterious effect for the newborn or parturient. In the absence of any observed complications, several teams began to use noradrenaline prophylactically in other surgery. However, no study has demonstrated its benefit, particularly the term of surgical complication in abdominal surgery. The objective of this work is to assess the preventive use of norepinephrine in major abdominal surgery on the occurrence of intraoperative hypotension, postoperative organ dysfunction and postoperative medical and surgical complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for major abdominal surgery (defined as surgery with a risk of cardiovascular complications of >1% and/or lasting more than 2 hours) with general anaesthesia.
* American Society of Anesthesiologists physical status (ASA-PS) score of ≥2.
* Age of ≥50 years and weighing more than 50 kg
* Written informed consent.

Exclusion Criteria:

* Emergency surgery.
* Untreated or uncontrolled hypertension (systolic blood pressure of >150 mm Hg), despite medication.
* Any acute cardiovascular event, including acute or decompensated heart failure or acute coronary syndrome.
* Patients with chronic kidney disease with a glomerular filtration rate of <30 ml.min-1/1.73 m2 or requiring renal replacement therapy for end-stage renal disease.
* Patients with severe hepatic failure (ASAT/ALAT of >2N, elevated bilirubin level, PT of <50%).
* Preoperative sepsis, septic shock.
* Preoperative norepinephrine infusion.
* Patients eligible for a surgical procedure under locoregional anaesthesia.
* Pregnancy.
* Known allergy to study treatment.
* Patients unable to give informed consent for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2025-11-29 (Actual)

PRIMARY OUTCOMES:
Variation of the of the Clavien Dindo surgical score between both groups | one month
  The Clavien-Dindo Classification
  The therapy used to correct a specific complication is the basis of this classification in order to rank a complication in an objective and reproducible manner.
  It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V). The introduction of the subclasses a and b allows a contraction of the classification into 5 grades (I, II, III, IV and V) depending on the size of the population observed or the of the focus of a study.
  Complications that have the potential for long-lasting disability after patient's discharge (e.g.: paralysis of a voice cord after thyroid surgery) are highlighted in the present classification by a suffix ("d" for disability). This suffix indicates that a follow-up is required to comprehensively evaluate the outcome and related long-term quality of life

SECONDARY OUTCOMES:
Variation of duration of hospital stay in days between both groups | one month
Length of intensive care unit stay | 1 month
length of postoperative care unit stay | 1 month
Postoperative renal function | at 48 hours
  Postoperative renal function assessed by the KDIGO score at 48 hours KDIGO (Kidney Disease: Improving Global Outcomes) stage 1 : Serum creatinine : 1.5-1.9 times baseline or ≥0.3 mg/dl (≥26.5μmol/l) increase stage 2 : Serum creatinine : 2.0-2.9 times baseline stage 3 : 3 times baseline or ≥4.0 mg/dl ( ≥353.6 μmol/l) increase stage 1 : Urine output : <0.5 ml/kg/h for 6-12 h stage 21 :Urine output : <0.5 ml/kg/h for ≥12 h stage 3 : Urine output : <0.3 ml/kg/h ≥24 h or anuria ≥12h
number of persistent circulatory shock | at 48 hours
  persistent circulatory shock defined by the use of vasoactive drugs beyond the 12th hour postoperatively
number of persistent circulatory shock | at 7 days
  persistent circulatory shock defined by the use of vasoactive drugs beyond the 12th hour postoperatively
number of persistent circulatory shock | at 1 month
  persistent circulatory shock defined by the use of vasoactive drugs beyond the 12th hour postoperatively
number of patients with cardiac rhythm disorder | at 1 month
  number of patients with cardiac rhythm disorder
number of patients with cardiac rhythm disorder | at 48 hours
  number of patients with cardiac rhythm disorder
number of patients with cardiac rhythm disorder | at 7 days
  number of patients with cardiac rhythm disorder
Number of patients with acute coronary syndrome | at 48 hours
  Number of patietns with acute coronary syndrome
Number of patients with acute coronary syndrome | at 1 month
  Number of patietns with acute coronary syndrome
Number of patients with acute coronary syndrome | at 7 days
  Number of patietns with acute coronary syndrome
Number of patients with Postoperative respiratory complications: respiratory infection | at 48 hours
  Number of patients with Postoperative respiratory complications: respiratory infection
Number of patients with Postoperative respiratory complications: respiratory infection | at 7 days
  Number of patients with Postoperative respiratory complications: respiratory infection
Number of patients with Postoperative respiratory complications: respiratory infection | at 1 month
  Number of patients with Postoperative respiratory complications: respiratory infection
Number of patients with Postoperative respiratory complications: atelectasis | at 1 month
  Number of patients with Postoperative respiratory complications: atelectasis
Number of patients with Postoperative respiratory complications: atelectasis | at 48 hours
  Number of patients with Postoperative respiratory complications: atelectasis
Number of patients with Postoperative respiratory complications: atelectasis | at 7 days
  Number of patients with Postoperative respiratory complications: atelectasis
Number of patients with Postoperative respiratory complications: oxygen support | at 7 days
  Number of patients with Postoperative respiratory complications: oxygen support
Number of patients with Postoperative respiratory complications: oxygen support | at 48 hours
  Number of patients with Postoperative respiratory complications: oxygen support
Number of patients with Postoperative respiratory complications: oxygen support | at 1 month
  Number of patients with Postoperative respiratory complications: oxygen support
Number of patients with Postoperative respiratory complications: mechanical ventilation | at 7 days
  Number of patients with Postoperative respiratory complications: mechanical ventilation
Number of patients with Postoperative respiratory complications: mechanical ventilation | at 48 hours
  Number of patients with Postoperative respiratory complications: mechanical ventilation
Number of patients with Postoperative respiratory complications: non-invasive ventilation | at 48 hours
  Number of patients with Postoperative respiratory complications: non-invasive ventilation
Number of patients with Postoperative respiratory complications: non-invasive ventilation | at 7 days
  Number of patients with Postoperative respiratory complications: non-invasive ventilation
Number of patients with Postoperative respiratory complications: non-invasive ventilation | at 1 month
  Number of patients with Postoperative respiratory complications: non-invasive ventilation
Number of patients with Postoperative respiratory complications: acute respiratory distress syndrome (ARDS) | at 48 hours
  Number of patients with Postoperative respiratory complications: acute respiratory distress syndrome (ARDS)
Number of patients with Postoperative respiratory complications: acute respiratory distress syndrome (ARDS) | at 7 days
  Number of patients with Postoperative respiratory complications: acute respiratory distress syndrome (ARDS)
Number of patients with Postoperative respiratory complications: acute respiratory distress syndrome (ARDS) | at 1 month
  Number of patients with Postoperative respiratory complications: acute respiratory distress syndrome (ARDS)
Number of patients with Infectious complications: sepsis | at 48 hours
  Number of patients with Infectious complications: sepsis
Number of patients with Infectious complications: sepsis | at 7 days
  Number of patients with Infectious complications: sepsis
Number of patients with Infectious complications: sepsis | at 1 month
  Number of patients with Infectious complications: sepsis
Number of patients with Infectious complications: sepsis shock | at 1 month
  Number of patients with Infectious complications: sepsis shock septic shock as defined in the international definitions (sepsis-related organ failure assessment score)
Number of patients with Infectious complications: sepsis shock | at 48 hours
  Number of patients with Infectious complications: sepsis shock septic shock as defined in the international definitions (sepsis-related organ failure assessment score)
Number of patients with Infectious complications: sepsis shock | at 7 days
  Number of patients with Infectious complications: sepsis shock septic shock as defined in the international definitions (sepsis-related organ failure assessment score)
Number of patients with Neurological complications: altered consciousness | at 7 days
  Number of patients with Neurological complications: altered consciousness
Number of patients with Neurological complications: altered consciousness | at 48 hours
  Number of patients with Neurological complications: altered consciousness
Number of patients with Neurological complications: altered consciousness | at 1 month
  Number of patients with Neurological complications: altered consciousness
Number of patients with Neurological complications: stroke | at 1 month
  Number of patients with Neurological complications: stroke
Number of patients with Neurological complications: stroke | at 48 hours
  Number of patients with Neurological complications: stroke
Number of patients with Neurological complications: stroke | at 7 days
  Number of patients with Neurological complications: stroke
Number of patients haematological complications: intraoperative blood loss | at 7 days
  Number of patients haematological complications: intraoperative blood loss
Number of patients haematological complications: intraoperative blood loss | at 48 hours
  Number of patients haematological complications: intraoperative blood loss
Number of patients haematological complications: blood transfusion and haemostasis disorder | at 48 hours
  Number of patients haematological complications: blood transfusion and haemostasis disorder
Number of patients haematological complications: blood transfusion and haemostasis disorder | at 7 days
  Number of patients haematological complications: blood transfusion and haemostasis disorder
Volume of intraoperative fluid therapy | at 48 hours
  Volume of intraoperative fluid therapy
Evaluation of the level of dependence in the activities of daily living | at 1 month post-discharge from the hospital
  Evaluation of the level of dependence in the activities of daily living : IADL scale The Lawton Instrumental Activities of Daily Living Scale (IADL) is an appropriate instrument to assess independent living skills There are eight domains of function measured with the Lawton IADL scale. Women are scored on all 8 areas of function; historically, for men, the areas of food preparation, housekeeping, laundering are excluded.
  Clients are scored according to their highest level of functioning in that category. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trocheris-Fumery O, Scetbon C, Flet T, Meynier J, Sellier M, Rumbach M, Badaoui R, Villeret L, Tarpin P, Abou-Arab O, Bar S, Dupont H. Evaluation of the early use of norepinephrine in major abdominal surgery on medical and surgical postoperative complications: study protocol for a randomised controlled trial (EPON STUDY). BMJ Open. 2024 Apr 29;14(4):e083606. doi: 10.1136/bmjopen-2023-083606. PMID 38684243